CLINICAL TRIAL: NCT06320418
Title: The Epigenetic Regulatory Role of P-element Induced Wimpy Testis (Piwi) Interacting RNA-
Brief Title: The Epigenetic Regulatory Role of P-element Induced Wimpy Testis (Piwi) Interacting RNA-823 (piR-823) in Ovarian Cancer Progression
Status: Active, not recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nadia Hamdy, professor of Biochemistry and molecular biology, Ain Shams University
Other Study IDs: RHDIRB2020110301REC#196
Record Dates: First submitted 2024-02-22; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Ovarian Cancer
Keywords: piR-823, Ovarian cancer, DNA methylation
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Ovarian fresh tissue samples were collected from the controls, and OC patients underwent surgical resection at the Department of Obstetrics and Gynecology, Ain Shams University. All resected tissue samples were stored at -20°C after adding RNA Stabilization Reagent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients group: A total of 39 female patients in their age range (13-75 years) diagnosed with primary malignant ovarian tumors were enrolled in the study. OC patients were a treatment-naïve Egyptian patients' cohort admitted to the Gynecology and Obstetrics Department or the Oncology Dept., Ain Shams University Hospitals, Cairo, Egypt. Ovarian cancer tissue samples were collected during surgical resection and confirmed by postoperative pathological examinations.
- Control group: A total of 17 normal ovarian tissue samples were collected from patients with benign uterine diseases, such as myoma, who underwent uterine and ovarian resection. The control's age range is 45-62 years

SUMMARY:
Ovarian cancer (OC) has one of the highest mortality rates for female malignant tumors, attributed to advanced cancer stages upon diagnosis as well as a high recurrence rate. Piwi-interacting RNA-823 (piR-823) is a single-stranded non-protein coding RNA (ncRNA) star molecule in epigenetics research. Extensive cellular regulatory functions and aberrant expression of piR-823 have been implicated in carcinogenesis. Therefore, the findings of piwi-ncRNA dysregulated-expression in OC Egyptian female patients' cohort could be employed as a potential novel mechanism for OC precision, a step toward ncRNA-precision

DETAILED DESCRIPTION:
1. Introduction Ovarian cancer (OC) represents one of the most aggressive female tumors worldwide and is the second most prevalent malignant tumor after breast cancer. In Egypt, OC represents the fourth most common female cancer. Current treatments become ineffective after several cycles of management due to the high recurrence rate, which is about 80-85%. Thus, it is urgent to explore novel targets for OC treatment [1]. OC represents a spectrum of diseases, not a single disease entity. Piwi-interacting RNA (piRNA) is a single-stranded non-coding RNA (ncRNA) with a nucleotide sequence of 23-35 that was discovered in mammalian germ cells. It has become a star molecule in non-coding RNA research due to its extensive cellular regulatory functions [3]. In recent years, many studies have found that piRNA is involved in tumor occurrence and development in many types of cancer, such as gastric cancer, liver cancer, lung cancer, breast cancer, and other cancers [4]. piR-52207 and piR-33733 participate in OC oncogenesis through involvement in numerous cell signaling pathways at the post-transcriptional level [5]. Nevertheless, the clinical significance and biological mechanisms of piRNAs in the progression of OC remain largely unknown. piR-823 was one of the first piRNAs recognized to be linked to malignancy and was identified in white blood cells, cancer cell lines, and blood plasma. piR-823 exhibits a pan-cancer expression pattern in various types of cancer, such as stomach, colon, breast, esophageal, liver, prostate, and renal cancer [6, 7]. More recently, piRNA-823 has been documented to be involved in tumorigenesis by regulating de novo DNA methylation and angiogenesis in multiple myeloma [3]. However, their functional mechanisms as well as their epigenetic regulatory role in OC have not been investigated Thus, investigating the regulatory role played by piR-823 could provide a way to explore the application of ncRNAs as a prognostic mechanism in OC, constituting a potential target for drug development RESEARCH OBJECTIVE(S) Investigate the expression level of piR-823 in OC tissue samples. Demonstrate the correlation between piR-823 and the progression of OC. Correlate piR-823 and OC clinicopathological characteristics
2. Subjects 2.1 Sample size and power of the study Sample size calculation is based on the previous study by (Jie Yin et al, 2017). Sample size estimation performed by G power* sample size online calculator (http://www.gpower.hhu.de/en.html), depending on two-sided confidence level 95%. The sample size to be able to reject the null hypothesis that the population means of the studied groups are equal with probability (power) (0.95) and type I error probability associated with this test of this null hypothesis is (0.05).

   2.2 Study design Case-controlled retrospective observational study, mono-center. 2.3 Institutional Review Board (IRB) statement The Research Ethics Committee of the Faculty of Pharmacy, Ain Shams University, granted ethical permission to conduct the study. All participants (controls or patients) were fully cognizant of the purpose of the study and signed a written, ethically-approved, informed consent (I·C) form. This study was conducted in accordance to the Declaration of Helsinki Guidelines approved in 2013 2.4 Study participant 2.4.1 Patients group A total of 39 female, their age range (13- 75 years), patients diagnosed with primary malignant ovarian tumor were enrolled in the study. OC patients were treatment-naïve Egyptian patients' cohort admitted to the Gynecology and Obstetrics Department or the Oncology Dept., Ain Shams University Hospitals, Cairo, Egypt. Ovarian cancer tissue samples were collected during surgical resection and confirmed by postoperative pathological examinations.

   2.4.2 Control group A total of 17 normal ovarian tissue samples were collected from patients with benign uterine diseases uterine such as myoma who underwent uterine and ovarian resection. Controls age range is 45-62 years For the patients' group (n = 39) a full history was recorded. Patient enrolled into the study If met the inclusion criteria and after giving their approval for participation in the study and signed the informed consent. Inclusion criteria; This study included newly diagnosed, untreated cases of histopathologically confirmed OC patients. Exclusion criteria; Individuals receiving chemotherapy, radiation, and patients with history of other cancer other than OC. Additionally, individuals with inadequate data or missing histopathological diagnoses.

   2.4.3. Patients' demographic data and pathological data Patients were either in the reproductive, premenopausal, or postmenopausal phase. The patients' demographic data including age, menopausal status, ascites, and the patient full history, retrieved from the patients' medical records collected from Ain Shams Hospitals in addition to the original pathology reports of the following data (tumor site, tumor size, tumor type, lymph node metastasis, distant metastasis, tumor stage, and tumor grade) were obtained from the Department of Pathology, Ain Shams Hospitals. OC histological staging made in accordance to the International Federation of Gynecology and Obstetrics (FIGO) criteria
3. Methods

3.1 in silico analysis Databases mining for targeting pathways and functional enrichment analysis in addition to Binding interaction predications 3.2 Tissue samples Ovarian fresh tissue samples were collected from the controls and OC patients underwent surgical resection at the Department of Obstetrics and Gynecology, Ain shams university. All resected tissue samples were stored at -20°C after adding RNA Stabilization Reagent (Qiagen, Hilden, Germany) 3.3 Total RNA extraction and quantification Using the miRNeasy Mini kit (Cat. No.217004; Qiagen, Hilden, Germany) according to the manufacturer's protocol, from tissue samples, Total RNA extraction was done. The isolated RNA was eluted in 40 μL of RNase-free water. Then, the isolated RNA quantified using NanoDrop® 1000 spectrophotometer (Thermo Scientific, Wilmington, DE, USA) the concentration and purity of all RNA samples were determined was stored at -80 °C in aliquots.

3.4 cDNA synthesis and measurement of piR-823 expression using qRT-PCR Total RNA will be reverse transcribed by miSCRIPT Kit (Qiagen, Hilden, Germany). Real-time PCR analysis subsequently performed using a miRcury LNA SYBR Green PCR Kit (Qiagen) as proposed by the manufacturer's instructions. The resulting cDNA was kept at -20 °C until quantification. qRT-PCR was used to measure the expression of the piR823 using the miRCURY LNA miRNA) endogenous control 3.5 cDNA synthesis and measurement of mRNA expression using qRT-PCR RevertAid First Strand cDNA Synthesis Kit (Thermo Scientific, Rockford, IL, USA) was used for cDNA synthesis according the manufacture instructions. qRT-PCR made using Power SYBR Green PCR Master Mix (Thermo Scientific, Rockford, IL, USA). GAPDH primer was used as endogenous control. The RNA relative expression was computed and normalized as fold change using the cycle threshold (Ct) method (2--ΔΔCt).

3.6 Statistical analysis

* Data will be collected, excel tabulated and tested for normality by Kolmogorov-Smirnov test.
* Between-group differences in age variability will be compared by the χ2 test and by analysis of variance for age variability. Multivariate logistic regression with adjustments for age will be used to show the association between selected piR-823 expression and OC risk.
* Normally distributed variables will be expressed as mean + (S.E.M) and analyzed using two samples independent t-test. Median (interquartile range) will be used to express nonparametric data, and subsequently analyzed using Mann Whitney U test.
* Pearson's Chi-square analysis or Fisher's exact test employed to compare the difference of categorical variables.
* For all analyses, a two-tailed P value of 0.05 or less considered statistically signiﬁcant

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients
* Untreated cases of patients
* Histopathologically confirmed OC patients

Exclusion Criteria:

* Individuals receiving chemotherapy, and radiation
* Patients with a history of other cancers other than ovarian cancer
* Individuals with inadequate data or missing histopathological diagnoses.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — study of ovarian cancer
Study Population: The patient enrolled in the study if they met the inclusion criteria and, after giving their approval for participation in the study, signed the informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Association of piR-823 expression with ovarian cancer progression | 18 months
  Investigating the expression of piR-823 in ovarian cancer tissue samples using qRT-PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Hamdy, PhD, Principal Investigator — faculty of pharmacy Ain Shams university
Locations (1):
- Faculty of Pharmacy, Ain Shams University, Advanced Biochemistry Research Lab, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] References [1] R. Jiang et al., "Inhibition of long non-coding RNA XIST upregulates microRNA-149-3p to repress OC cell progression," Cell Death Dis., vol. 12, no. 2, p. 145, Feb. 2021, doi: 10.1038/s41419-020-03358-0. [3] E. Lee, N. A. Lokman, et al. "A Comprehensive Molecular and Clinical Analysis of the piRNA Pathway Genes in OC," Cancers (Basel)., vol. 13, no. 1, p. 4, Dec. 2020, doi: 10.3390/cancers13010004. [4] K. Wang, T. Wang, X. Gao, X. Chen, F. Wang, and L. Zhou, "Emerging functions of piwi-interacting RNAs in diseases," J. Cell. Mol. Med., vol. 25, no. 11, pp. 4893-4901, Jun. 2021, doi: 10.1111/jcmm.16466. [5] G. Singh, J. Roy, P. Rout, and B. Mallick, "Genome-wide profiling of the PIWI-interacting RNA-mRNA regulatory networks in epithelial OCs," PLoS One, vol. 13, no. 1, p. e0190485, Jan. 2018, doi: 10.1371/journal.pone.0190485. [6] N. A. Sabbah et al., "piRNA-823 Is a Unique Potential Diagnostic Non-Invasive Biomarker in Colorectal Cancer Patients," Genes (Basel)., vol. 12, no. 4, p. 598, Apr. 2021, doi: 10.3390/genes12040598. [7] J.-F. Su et al., "piR-823 demonstrates tumor oncogenic activity in esophageal squamous cell carcinoma through DNA methylation induction via DNA methyltransferase 3B," Pathol. - Res. Pract., vol. 216, no. 4, p. 152848, Apr. 2020, doi: 10.1016/j.prp.2020.152848.